CLINICAL TRIAL: NCT06990048
Title: The Long-Term EVAR Assessment and Follow-Up (LEAF) Study for the AFX2 System
Acronym: LEAF
Status: Recruiting | Type: Observational
Sponsor: Endologix (Industry)
Collaborators: Fivos (Unknown)
Responsible Party: Sponsor
Other Study IDs: CP-0024
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: AFX2 System — The AFX2 System comprises of the following:
  AFX2 Bifurcated Endograft System and delivery system AFX Vela Proxmal Endograft System and delivery system AFX Stand Alone Endograft System and delivery system

SUMMARY:
This is an observational, retrospective, multicenter study to evaluate the performance of the AFX2 System using real world evidence from VQI-VISION.

DETAILED DESCRIPTION:
Evaluate the clinical performance of the AFX2 System patients against other commercially available EVAR devices and evaluate the Type III endoleak occurrence in AFX2 System patients through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients implanted with the AFX2 System or the 3 most commonly used comparator devices who underwent EVAR as their first abdominal aortic aneurysm repair in the VQI EVAR registry will be included in this study.

Exclusion Criteria:

* Ruptured AAA repair with the AFX2 or comparator device
* Patients with AFX2 in AFX relining, or relined comparator grafts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 20,000 patient data will be extracted from approximately 900 sites participating in the VQI EVAR registry in the US. A minimum of 2000 AFX2 System patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rates of AAA Rupture, Reintervention and Mortality | 5 Years
  Rate of the composite of AAA rupture, aortic-related reintervention, and morality through 5 years.
Incidence of Endoleak | 5 Years
  Cummulative incidence of Type III endoleaks at 5 years.

SECONDARY OUTCOMES:
Long Term Safety | 10 Years
  Rates of AAA rupture, aoritic-related reintervention, mortality, aneurysm related mortality, rate of imaging with CT, presence of untreated asymptomatic Type III endoleaks, occurrence of sac shrinkage, stability, and expansion >5mm in diameter, and limb occlusion at 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- The Dartmouth Institute, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No